CLINICAL TRIAL: NCT00635700
Title: Ziprasidone vs Placebo in the Prevention of Psychosis Among Symptomatic Adolescents and Young Adults at Prodromal Risk
Brief Title: Ziprasidone in the Psychosis Prodrome
Acronym: ZIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0801003386; IIR GA1281GE
Record Dates: First submitted 2008-03-06; First posted 2008-03-14 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Psychosis Prodrome
Keywords: psychosis; schizophrenia; prodrome; ziprasidone; placebo
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ziprasidone (Experimental): Patients will be treated with Ziprasidone for 6 months
  Interventions: Drug: ziprasidone
- Placebo (Placebo Comparator): Patients will be treated with placebo for 6 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ziprasidone — 20-160 mg/d
  Other Names: Geodon
  Arms: Ziprasidone
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
This study aims to determine whether ziprasidone is superior to placebo over 24 weeks for patients with the psychosis prodrome.

ELIGIBILITY:
Inclusion Criteria:

* Structured Interview for Psychosis-risk Syndromes criteria for Clinical High Risk for Psychosis
* clinically referred

Exclusion Criteria:

* prolonged corrected QT interval
* history of syncope

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2008-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Woods, MD, Principal Investigator — Yale University
Locations (11):
- United States (10):
  - University of California at San Diego, La Jolla, California
  - University of California at Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Beth Israel Deaconess Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Wayne State University School of Medicine, Detroit, Michigan
  - North Shore, Long Island Jewish Health System, Glen Oaks, New York
  - University of North Carolina, Chapel Hill, North Carolina
- University of Calgary, Calgary, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ziprasidone | Placebo
Started | 24 | 27
Completed | 9 | 13
Not Completed | 15 | 14

BASELINE CHARACTERISTICS:
Population: Of 51 patients randomized, 27 were assigned to placebo and 24 to ziprasidone. One case allocated to ziprasidone was never dispensed study medication and was removed from analysis per protocol, leaving 23.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone | Placebo | Total
Number analyzed (Participants) | 23 | 27 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.9 (4.7) | 22.6 (3.7) | 22.3 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 13 | 19 | 32
Region of Enrollment [Number; unit: participants]
  United States | 23 | 27 | 50

OUTCOME MEASURES:

1. Primary Outcome: Conversion to Psychosis
Description: Conversion to psychosis according to the Structured Interview for Psychosis-risk Syndromes (SIPS) require psychotic symptom severity ratings in the frankly psychotic range, along with meeting persistence or urgency criteria.
Time Frame: 6 months
Population: In another case assigned to active ziprasidone, ratings conducted at a follow-up conversion visit suggested retrospectively that the patient had been already psychotic prior to enrollment. The study's blinded DSMB was consulted, and in a split 4-2 vote recommended retaining the patient as randomized in the primary analysis.
Measure: Number; unit: participants
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 23 | 27
participants | 1 | 2

2. Secondary Outcome: Change in Scale of Psychosis-risk Symptoms Total Score
Description: The Scale of Psychosis-risk Symptoms, a 19-item scale with items scored 0-6. Positive Symptom scores on the SOPS in the 1 to 2 range are considered non-prodromal. Scores of 6 are considered psychotic. Scores in the 3 to 5 range are considered at the clinical high risk level. Minimum value 0. Maximum value 114. Higher score means worse outcome.
Time Frame: baseline and 8 weeks
Population: All subjects who received allocated intervention
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 23 | 27
scores on a scale | -0.271 [-0.693 to 0.152] | 0 [0 to 0]

ADVERSE EVENTS:
Arm/Group | Ziprasidone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 1/24 | 2/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ziprasidone (N=24) | Placebo (N=27)
EKG abnormalities (Cardiac disorders) | 1 (1) | 2 (2) — Any emergent EKG abnormality including QTcF prolongation > 460 msec, or 15% of baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No